CLINICAL TRIAL: NCT00729885
Title: Visual Feedback Goggle For The Treatment Of Benign Paroxysmal Positional Vertigo in a Randomized Single-Blind Study
Brief Title: Visual Feedback Goggle for Positional Vertigo Treatment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vertigone Inc. (Industry)
Responsible Party: Philip F. Anthony, MD, Vertigone, Inc
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: V200601
Record Dates: First submitted 2008-08-01; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Positional Vertigo; Vertigo
Keywords: Vertigo; Benign Paroxysmal Positional Vertigo; BPPV; Positional Vertigo
MeSH Terms: conditions — Vertigo; Benign Paroxysmal Positional Vertigo | interventions — Eye Protective Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Goggle I (Experimental): Optimized Goggle
  Interventions: Device: Optimized Goggle
- 2 Google II (Sham Comparator): Goggle with 20 Degree error
  Interventions: Device: Goggle with 20 degree error

INTERVENTIONS:
Device: Goggle with 20 degree error — The Vertigone Goggle is modified such that the head positions and visual feedback indicators are offset 20° from the classic Epley positions.
  Arms: 2 Google II
Device: Optimized Goggle — The classic Epley maneuver involves 3 head positions: 1) the patient supine, the neck is extended 20°and the head turned 45° towards the affected ear, 2) the patient rotates his head 90° to the contralateral side, with the final head position 45° from vertical, 3) the patient turns his head 135° towards the floor on the contralateral side. For the classic Epley maneuver, the goggle coach ball markings will be set for correct positioning.
  Arms: 1 Goggle I

SUMMARY:
Benign Paroxysmal Positional Vertigo (BPPV) is one of the most common causes of vertigo and the most common vestibular disorder of the inner ear. BPPV is the result of small free-floating particles (canaliths) in the posterior semicircular canals where they aggravate the sensory apparatus and induce sudden and severe attacks of vertigo when the head is turned into certain positions.

The treatment of BPPV was revolutionized by the introduction of the Epley maneuver, a sequence of head movements that use gravity to reposition the canaliths within the inner ear. The Epley maneuver provides prompt relief from vertigo in approximately 80% of patients.

The innovation, the Vertigone goggle, provides both physician and patient with visual feedback to guide them through an accurate Epley maneuver. This changes the current treatment paradigm for BPPV, greatly increasing the availability of the maneuver to non-specialist physicians, nurse practitioners, physician's assistants and physical therapists. The device is designed so that the patient with recurrent vertigo can use the goggle to treat BPPV at home. The goggle is currently a pre-market prototype.

The hypothesis for the study is that accuracy in the performance of the Epley maneuver correlates with improved clinical resolution of vertigo in BPPV patients. If the hypothesis is true, then there is a clear case for the utility of the visual feedback provided by the VertiGONE goggle in performing the maneuver.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30-80
* Old patients (more than one year since first symptom)or new patients(more than 3 months duration of symptoms) diagnosed by physicians with Benign Paroxysmal Positional Vertigo (BPPV)
* Must have good neck flexibility to perform the movements of the Epley maneuver
* Subject is willing and able to provide written informed consent
* Subject is willing to remain in the clinic for the treatment and follow-up visits

Exclusion Criteria:

* Age < 30 or Age > 80
* Can not perform the movements of the Epley maneuver
* No informed consent form
* Not willing to remain in the clinic for the treatment and follow-up visits

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Symptom Relief Speed (SRS): defined as the number of days post-treatment until dizziness symptoms improve to category 5 (70-100% improvement from baseline). | This endpoint will be measured twice: once following the baseline visit and again following the subsequent visit and treatment.
Symptom Relief Completeness (SRC): defined as the highest level (on the ordinal scale) of improvement attained during the allotted seven-day time period. | This endpoint will also be measured twice, in the same manner as was SRS.

CONTACTS AND LOCATIONS:
Overall Officials: Philip F Anthony, MD, Principal Investigator — Vertigone Inc.
Locations (3):
- United States (3):
  - Jay Farrior, MD, Tampa, Florida
  - Debra Cooke, PH.D., Kansas City, Missouri
  - Mitchell Schwaber, MD, Nashville, Tennessee

REFERENCES:
- See also: Vertigone, Inc. 901 Hemphill Street, Fort Worth, Texas 76104 — http://www.vertigone.com